CLINICAL TRIAL: NCT03438695
Title: Total Motorized Spiral Enteroscopy Trial
Acronym: TMSET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Evangelisches Krankenhaus Düsseldorf (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TMSET 1.0
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Small Bowel Disease
Keywords: endoscopy, motorized spiral enteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Motorized Spiral Enteroscopy (Experimental): Patients with indication for total enteroscopy. day1: anterograde motorized spiral enteroscopy, day 2: retrograde motorized spiral enteroscopy
  Interventions: Procedure: Motorized Spiral Enteroscopy

INTERVENTIONS:
Procedure: Motorized Spiral Enteroscopy — Motorized Spiral endoscope will be inserted and advanced with the assistance of motorized clockwise spiral rotation, After reaching the cecum or if no further advancement of the endoscope can be achieved depth of insertion required for patient treatment or diagnosis, the endoscope will be withdrawn using motorized counter-clockwise spiral rotation, also controlled by the foot pedal. If no total enteroscopy was achieved, a submucosal ink dye injection is performed as an endoscopically visible marker of the maximum insertion depth. A retrograde peranal enteroscopy is then performed on one of the following days.

SUMMARY:
Study design Prospective bicentric non-controlled clinical trial

Study purpose

- to evaluate the efficacy and safety of Novel Motorized Spiral Enteroscopy (NMSE) for total enteroscopy in patients with suspected small bowel diseases with an indication for direct visualization of the entire small bowel

Primary objective

Rate of total enteroscopy by means of NMSE with:

1. a complete anterograde approach
2. or a combined anterograde and retrograde approach

Secondary objectives

* Procedural success of anterograde and retrograde approach
* Procedural time (minutes)
* Depth of maximum insertion (cm)
* Diagnostic yield
* Therapeutic yield
* Adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients with small bowel disease with an indication for a total enteroscopy, e.g.:
* Overt obscure gastrointestinal bleeding or obscure gastrointestinal bleeding or indeterminate iron-deficiency anaemia and positive Video capsule endoscopy (VCE) or negative VCE in patients who have ongoing bleeding shown by overt bleeding or continued need for blood transfusions
* Abdominal pain or chronic diarrhoea with positive findings of small bowel imaging examinations
* Noncontributory ileocolonoscopy and suspicion of Crohn's disease on small-bowel cross-sectional imaging modalities or small-bowel capsule endoscopy
* Further evaluation of known Crohn's disease or therapeutic indications in Crohn's disease
* Large polyps (>10-15mm) in the jejunum and ileum discovered by radiological examination or small-bowel capsule endoscopy in patients with Peutz-Jeghers syndrome
* Nonresponsive or refractory coeliac disease

Exclusion Criteria:

* - Age under 18 years
* Health status American Society of Anesthesists Classification (ASA) 4
* Pregnancy
* Coagulopathy (INR≥2.0, Platelets < 70/nl)
* Taking anti-platelet agents or anticoagulants (other than aspirin) within last 7 days
* Any medical contraindication to standard enteroscopy
* Presence of any intraluminal or extraluminal foreign body in the abdominal cavity
* Any prior gastric, small bowel or colonic surgery, or implantable devices in these locations (cardiac pacemakers and non-abdominal implants are acceptable)
* Known or suspected bowel obstruction or stenosis or history of bowel obstruction
* Known coagulation disorder
* Known or suspected esophageal stricture or Schatzki ring
* Known gastric or esophageal varices
* Suspected perforation of the GI tract
* Known or suspected colonic or ileocecal valve (ICV) stricture
* Inability to tolerate sedation or general anesthesia for any reason
* Inability to tolerate endotracheal intubation
* Absence of a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-21 (Estimated); Primary Completion 2019-02-21 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of total enteroscopy by Motorized Spiral Enteroscopy | 2 days
  Total enteroscopy by:
  1. a complete anterograde approach
  2. or a combined anterograde and retrograde approach

SECONDARY OUTCOMES:
Procedural Success Rate | 2 days
  of anterograde and retrograde approach
Procedural time | 2 days
  of anterograde and retrograde approach
Depth of maximum insertion to the small bowel | 2 days
  anterograde and retrograde
Diagnostic yield | 2 days
  anterograde and retrograde
Therapeutic yield | 2 days
  anterograde and retrograde
Adverse events | 3 days
  anterograde and retrograde, serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Beyna, MD, Study Chair — EVK Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beyna T, Arvanitakis M, Schneider M, Gerges C, Hoellerich J, Deviere J, Neuhaus H. Total motorized spiral enteroscopy: first prospective clinical feasibility trial. Gastrointest Endosc. 2021 Jun;93(6):1362-1370. doi: 10.1016/j.gie.2020.10.028. Epub 2020 Nov 2. PMID 33144239